CLINICAL TRIAL: NCT06417060
Title: THE IMPACT OF CAUDAL BLOCK ANESTHESIA ON POSTOPERATIVE COMPLICATIONS IN DISTAL HYPOSPADIAS SURGERY: A MULTI-CENTER RANDOMIZED CONTROLLED TRIAL
Brief Title: Caudal Anesthesia Versus Local Anesthesia in Hypospadias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmi Kadıoğlu Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Azizoğlu, MD, Necmi Kadıoğlu Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hypospadias; Hypospadias, Coronal; Caudal Anesthesia; Children
Keywords: Hypospadias; Caudal anesthesia; Urethrocutanous fistula
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Experimental): Anesthesia will be administered via inhalation induction with air/nitrous oxide and sevoflurane, followed by an injection of 0.25% bupivacaine (1 mL/kg) without epinephrine into the caudal canal, which is the sacral portion of the spinal canal.
  Interventions: Drug: Caudal block anesthesia
- Dorsal Penile Block Anesthesia (Sham Comparator): Anesthesia will be administered using an inhalation induction method with air/nitrous oxide and sevoflurane, followed by the injection of 0.25% bupivacaine without epinephrine into the dorsal part of the penis.
  Interventions: Drug: Dorsal penile block anesthesia

INTERVENTIONS:
Drug: Caudal block anesthesia — Anesthesia will be administered via inhalation induction with air/nitrous oxide and sevoflurane, followed by an injection of 0.25% bupivacaine (1 mL/kg) without epinephrine into the caudal canal, which is the sacral portion of the spinal canal.
  Arms: Caudal block
Drug: Dorsal penile block anesthesia — Anesthesia will be administered using an inhalation induction method with air/nitrous oxide and sevoflurane, followed by the injection of 0.25% bupivacaine without epinephrine into the dorsal part of the penis.
  Arms: Dorsal Penile Block Anesthesia

SUMMARY:
Hypospadias is among the most common congenital genital malformations in boys and is typically treated through surgical intervention. During pediatric urological surgery, caudal anesthesia, also known as a caudal block, is frequently employed as a regional anesthetic technique. It has proven to be a safe and effective anesthetic approach in children, with a low rate of anesthesia-related complications. However, despite the low incidence of complications directly associated with the caudal block, there is limited and inconclusive evidence regarding its impact on surgical complications. Therefore, this randomized controlled superiority trial aims to evaluate whether the use of caudal anesthesia, compared to the dorsal penile block, is associated with an increased incidence of urethrocutaneous fistulas and glans dehiscence following hypospadias repair.

DETAILED DESCRIPTION:
The rationale for conducting a comprehensive study arises from the limitations inherent in existing literature, primarily due to selection bias and the retrospective nature of current evidence, which fails to clarify whether caudal blocks lead to higher complication rates after hypospadias repair. To fill this knowledge gap and address the clinical uncertainty surrounding this issue, the only effective approach is to randomly assign patients undergoing hypospadias repair to receive either caudal or penile block anesthesia. The purpose of this pilot study is to evaluate the feasibility of a definitive trial and identify any methodological issues that must be resolved before committing significant resources to a full-scale study.

This pilot study will assess the feasibility of conducting a large, definitive, parallel-group, randomized controlled trial (RCT) to determine whether a dorsal penile block results in fewer postoperative complications than a caudal block in boys aged 6 to 48 months undergoing hypospadias repair.

Hypospadias repair will be performed under standardized analgesic administration, and participants may receive fentanyl (1-3 mcg/kg) at the anesthesiologist's discretion. Anesthesia will be induced via inhalation of air/nitrous oxide and sevoflurane. Based on a randomized allocation, patients will receive either a caudal anesthetic block (0.25% bupivacaine, 1 ml/kg, up to a maximum of 10 ml) or a dorsal penile block (bupivacaine without epinephrine, 10-20 ml/kg). All patients will receive antiemetic prophylaxis with dexamethasone (150 mcg/kg), ondansetron (50 mcg/kg), acetaminophen suppository (40 mg/kg), and intravenous morphine (0.02-0.1 mg/kg).

At discharge, patients will be prescribed oral morphine (0.2 mg/kg) every 4 hours as needed, Ditropan (0.2 mg/kg) every 12 hours as needed, Tylenol (15 mg/kg per dose) every 4 hours, or ibuprofen (10 mg/kg per dose) every 6 hours. Parents will administer these medications at their discretion. Trimethoprim (2 mg/kg) will also be prescribed until catheter removal.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 48 months
* Distal hypospadias
* Acceptance of participation

Exclusion Criteria:

* Midpenil hypospadias
* Proximal hypospadias
* Prior surgery
* Comorbidity (diabetes, hypertention, cardiac pathology)

Ages: 6 Months to 48 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-08-29 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative complication rate | 1 year
  A urethrocutaneous fistula (UCF) is characterized by an abnormal connection between the reconstructed urethra and the skin, situated between the original meatus and the tip of the penis. Glans dehiscence refers to the complete separation of the glans wings, which may or may not be connected by a strip of skin.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoğlu, Principal Investigator — Necmi Kadıoğlu State Hospital
Locations (3):
- Ss. Cyril and Methodius University in Skopje, Pediatric Surgery, Skopje, Macedonia, the former Yugoslav Republic of North Macedonia, Skopje, North Macedonia
- Ao Gk Medsi, Moscow, Russia
- Necmi Kadioglu Esenyurt State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No